CLINICAL TRIAL: NCT04777344
Title: Clinical Effort Against Smoke Exposure in Cystic Fibrosis (CEASE-CF)
Brief Title: Clinical Effort Against Smoke Exposure in Cystic Fibrosis
Acronym: CEASE-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Gabriela R Oates, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300006654
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis
Keywords: caregivers; tobacco; smoke exposure
MeSH Terms: conditions — Cystic Fibrosis | interventions — Methods

STUDY DESIGN:
Intervention Model Description: single-center, randomized, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive the multi-component intervention (counseling with intake assessment, follow-up, help obtaining nicotine replacement therapy, and CF-specific smoke exposure education)
  Interventions: Behavioral: Tobacco Treatment Specialist (TTS) intervention
- Control group (No Intervention): The control group will receive usual care plus CF-specific smoke exposure education.

INTERVENTIONS:
Behavioral: Tobacco Treatment Specialist (TTS) intervention — A trained Tobacco Treatment specialist (TTS) embedded in the multi-disciplinary CF care team will provide tobacco use counseling to smoking caregivers of children with CF.
  Arms: Intervention group

SUMMARY:
The study will test the feasibility, acceptability, and preliminary efficacy of a multi-component smoking cessation intervention tailored to the needs of caregivers of children with CF and delivered in clinical settings as part of routine CF care. The ultimate goal of this effort is to reduce the exposure of children and adolescents with CF to tobacco smoke.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label study to test the feasibility and acceptability (primary outcomes) and preliminary efficacy (secondary outcome) of a multi-component smoking-cessation intervention delivered by a tobacco treatment specialist (TTS) integrated in the multidisciplinary CF care team.

The intervention will be tested in a two-group design with a 2:1 allocation. Participants (dyads of caregiver/CF child) will be randomized to either intervention or control group. The intervention group (N=24) will receive the multi-component intervention (intake assessment, follow-up, help with obtaining nicotine replacement therapy, and CF-specific smoke exposure education). The control group (N=12) will receive usual care plus CF-specific smoke exposure education.

ELIGIBILITY:
Inclusion Criteria:

* Adult familial caregiver of a child with CF aged <18 years
* Speak English
* Report smoking at least 1 cigarette in the previous week
* Not enrolled in a smoking cessation program

Exclusion Criteria:

* Do not report smoking at least 1 cigarette in the previous week
* Currently enrolled in a smoking cessation program.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | 6 months
  Participant drop-out rates and time added to the clinical encounter
Intervention acceptability | 6 months
  Proportion of caregivers who accepted participation; Participant and provider satisfaction with the intervention on a 1-5 Likert scale; Perceived effectiveness of the intervention on a 1-5 Likert scale

SECONDARY OUTCOMES:
Self-reported caregiver cessation | 6 months
  7-day point prevalence of abstinence measured at 1, 3, and 6 months; Number of cigarettes smoked in the past 7 days, measured at 1, 3, and 6 months
Child smoke exposure | 6 months
  Biochemically verified with a hair nicotine sample at baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niranjan SJ, Woods BM, Coleman E, Geurs R, Ladores-Barrett S, Oates GR. "It Was All Tailored Around Me": Qualitative Evaluation of Clinical Effort Against Smoke Exposure in Cystic Fibrosis (CEASE-CF). Pediatr Pulmonol. 2026 Feb;61(2):e71496. doi: 10.1002/ppul.71496. PMID 41657041